CLINICAL TRIAL: NCT03192332
Title: Solitaire™ With the Intention For Thrombectomy Plus Intravenous t-PA Versus DIRECT Solitaire™ Stent-retriever Thrombectomy in Acute Anterior Circulation Stroke
Brief Title: Bridging Thrombolysis Versus Direct Mechanical Thrombectomy in Acute Ischemic Stroke
Acronym: SWIFT DIRECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-00974
Record Dates: First submitted 2017-06-12; First posted 2017-06-20 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Ischemic Stroke
Keywords: Intravenous thrombolysis; Endovascular treatment; Mechanical thrombectomy; Bridging thrombolysis; Acute ischemic stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, open label, blinded endpoint (PROBE)
Who Masked: Outcomes Assessor
Masking Description: Assessment of the primary outcome will be performed by an independent and blinded person.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Direct mechanical thrombectomy (Experimental): Treatment with direct mechanical thrombectomy with a commercially available stent-retriever revascularization device of the Solitaire™ type.
  Interventions: Device: Stent-retriever thrombectomy with revascularization device of the Solitaire™ type
- Combined intravenous thrombolysis and mechanical thrombectomy (Active Comparator): Treatment with intravenous thrombolysis with recombinant tissue-type plasminogen activator (IV t-PA) followed by mechanical thrombectomy with a commercially available stent-retriever revascularization device of the Solitaire™ type.
  Interventions: Device: Stent-retriever thrombectomy with revascularization device of the Solitaire™ type; Drug: Intravenous thrombolysis with recombinant tissue-type plasminogen activator (IV t-PA)

INTERVENTIONS:
Device: Stent-retriever thrombectomy with revascularization device of the Solitaire™ type — Mechanical thrombectomy with a stent-retriever revascularization device
Drug: Intravenous thrombolysis with recombinant tissue-type plasminogen activator (IV t-PA) — Bridging thrombolysis (IV t-PA plus mechanical thrombectomy) according to current European and North American stroke guidelines.
  Arms: Combined intravenous thrombolysis and mechanical thrombectomy

SUMMARY:
Intravenous thrombolysis with recombinant tissue-type plasminogen activator (IV t-PA) has been the only proven therapy for acute ischemic stroke (AIS) for almost 20 years. Whether IV t-PA prior to endovascular clot retrieval is beneficial for AIS patients with a proximal vessel occlusion in the anterior circulation has currently become a matter of debate and is a relevant unanswered question in clinical practice.

The main objective is to determine whether subjects experiencing an AIS due to large intracranial vessel occlusion in the anterior circulation will have non-inferior functional outcome at 90 days when treated with direct mechanical thrombectomy (MT) compared to subjects treated with combined IV t-PA and MT.

The secondary objectives are to study causes of mortality, dependency and quality of life in these AIS patients.

DETAILED DESCRIPTION:
Intravenous thrombolysis with recombinant tissue-type plasminogen activator (IV t-PA) has been the only proven therapy for acute ischemic stroke (AIS) for almost 20 years. Since December 2014 a new era in acute stroke treatment has begun: randomized controlled studies have consistently shown that endovascular clot retrieval in addition to best medical treatment (± IV t-PA) improves outcome in acute anterior circulation stroke patients with proximal vessel occlusion compared to best medical treatment alone. Whether pre-treatment with IV t-PA prior to endovascular clot retrieval is beneficial has now become a matter of debate. A pooled analysis of 5 RCTs (MR CLEAN, SWIFT-PRIME, EXTEND IA, ESCAPE and REVASCAT) suggested that the treatment effect size of MT does not differ between patients receiving intravenous thrombolysis (IVT) and those treated with MT alone (p interaction: 0.4311). Besides post-hoc RCT analyses, there are a myriad of observational studies reporting on rates of successful reperfusion and functional outcome stratified according to IV t-PA pretreatment status. There is evidence that reperfusion rates after IV t-PA in patients with occlusions of the internal carotid artery and the main stem of the middle cerebral artery are low, but may reach more than 80% after mechanical thrombectomy (MT). Therefore the most important factor for vessel recanalization, which is linked with favorable outcome, is MT.

No randomized controlled trial has ever assessed whether direct MT in patients with AIS is equally effective as MT in combination with IV t-PA (bridging thrombolysis). In a patient-level pooled analysis of five randomized controlled studies (HERMES collaboration) similar rates of functional independence and mortality at 90 days were observed between patients who received IV t-PA+MT and those who received direct MT. However, patients in the direct MT group had contraindications for IV t-PA. Two larger studies based on registries compared the outcome of patients after bridging thrombolysis with direct MT in patients eligible for IV t-PA. In both studies, the outcome of patients after bridging thrombolysis and direct MT was similar. For these reasons the investigators hypothesize that immediate and direct MT is not inferior and might even be superior to bridging thrombolysis in patients directly referred to a stroke center with rapid access to endovascular procedures.

In this trial all commercially available stent-retriever revascularization devices manufactured by Medtronic (e.g. Solitaire™) will be used as tool for direct MT. The investigators aim to provide conclusive information on the efficacy and safety of direct MT, in comparison with bridging thrombolysis.

If direct MT in patients with AIS would not be inferior to bridging thrombolysis, the organization of acute stroke management would change essentially. Direct MT would then be the therapy of choice in stroke centers with endovascular facilities. Furthermore, this trial could have an impact on healthcare guidelines and costs. However, this trial does not address the question, whether patients arriving in stroke units with no endovascular facilities should be pre-treated with IV t-PA or whether they should directly be referred to stroke centers with endovascular facilities.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent as documented by signature
2. Age ≥ 18
3. Clinical signs consistent with an acute ischemic stroke
4. Neurological deficit with a NIHSS of ≥ 5 and < 30 (deficits judged to be clearly disabling at presentation)
5. Patient is eligible for intravenous thrombolysis
6. Patient is eligible for endovascular treatment
7. Randomization no later than 4 hours 15 minutes after stroke symptom onset and initiation of IV t-PA must be started within 4 hours 30 minutes of stroke symptoms onset (onset time is measured from the time when the subject was last seen well)
8. Occlusion (TICI 0-1) of the intracranial internal carotid artery (ICA), the M1 segment of the middle cerebral artery (MCA), or both confirmed by CT or MR angiography, accessible for MT
9. Core-infarct volume of Alberta Stroke Program Early CT Score (ASPECTS) greater than or equal to 4 (≥ 4) based on baseline CT or MR imaging (MRI) (a region has to have diffusion abnormality in 20% or more of its volume to be considered MR-ASPECTS positive)

Exclusion Criteria:

1. Acute intracranial hemorrhage
2. Any contraindication for IV t-PA
3. Pre-treatment with IV t-PA
4. In-hospital stroke
5. Pregnancy or lactating women. A negative pregnancy test before randomization is required for all women with child-bearing potential.
6. Known (serious) sensitivity to radiographic contrast agents, nickel, titanium metals, or their alloys
7. Known current participation in a clinical trial (investigational drug or medical device)
8. Renal insufficiency as defined by a serum creatinine > 2.0 mg/dl (or 176.8 µmol/l) or glomerular filtration rate (GFR) < 30 mL/min or requirement for hemodialysis or peritoneal dialysis
9. Severe comorbid condition with life expectancy less than 90 days at baseline
10. Known advanced dementia or significant pre-stroke disability (mRS score of ≥2)
11. Foreseeable difficulties in follow-up due to geographic reasons (e.g. patients living abroad)
12. Comorbid disease or condition that would confound the neurological and functional evaluations or compromise survival or ability to complete follow-up assessments.
13. Subject currently uses or has a recent history of illicit drug(s) or abuses alcohol (defined as regular or daily consumption of more than four alcoholic drinks per day).
14. Known history of arterial tortuosity, pre-existing stent, other arterial disease and/or known disease at the femoral access site that would prevent the device from reaching the target vessel and/or preclude safe recovery after MT
15. Radiological confirmed evidence of mass effect or intracranial tumor (except small meningioma)
16. Radiological confirmed evidence of cerebral vasculitis
17. CTA or MRA evidence of carotid artery dissection
18. Evidence of additional distal intracranial vessel occlusion in another territory (i.e. A2 segment of anterior cerebral artery or M3, M4 segment of MCA) on initial NCCT/MRI or CTA/MRA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2021-08-11 (Actual)

PRIMARY OUTCOMES:
Score in modified Rankin Scale (mRS) | 90 days after randomization

SECONDARY OUTCOMES:
Mortality | 90 days after randomization
Modified Rankin Scale (mRS) shift analysis | day 0 and 90 days after randomization
National Institute of Health Score Scale (NIHSS) | day 0 and day 1 after randomization
Thrombolysis in Cerebral Infarction (TICI) scale | day 0 and day 1 after randomization
Serious adverse events | day 0 until 90 days after randomization
Intracranial hemorrhage | day 1 after randomization
Quality of life assessed by questionnaire | 90 days after randomization
Overall costs incurred during hospitalisation | 90 days after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Urs Fischer, Prof. Dr., Principal Investigator — Dept. of Neurology, Inselspital Bern; Jan Gralla, Prof. Dr., Principal Investigator — Dept. of Neuroradiology, Inselspital Bern
Locations (48):
- Austria (2):
  - Keppler Universitätsklinikum, Linz, Upper Austria
  - Medical University of Innsbruck, Innsbruck
- Canada (4):
  - University of Calgary, Alberta Health Services, Calgary
  - Mc Gill University, Montreal
  - Royal University Hospital, University of Saskatchewan, Saskatoon
  - Toronto Western Hospital, Toronto
- Helsinki University Hospital, Helsinki, Finland
- France (19):
  - Hôpital Cavale Blanche CHU Brest, Brest, Finistère
  - CHU de Reims, Reims, Marne
  - CHU de Clermont-Ferrand, Clermont-Ferrand, Puy-de-Dôme
  - CHU de Bordeaux, Bordeaux
  - CHU de Caen Normandie, Caen
  - CHU de Lille, Lille
  - CHU de Limoges, Limoges
  - Hospices Civils de Lyon, Lyon
  - CHU de Montpellier, Montpellier
  - CHRU Nancy, Nancy
  - CHU de Nantes, Nantes
  - Hôpital Bicêtre, Paris
  - GHU Paris Psychiatrie et Neurosciences, Sainte Anne, Paris
  - Fondation Ophtalmologique A. de Rothschild, Paris
  - CHU Rouen Normandie, Rouen
  - CHRU Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse
  - CHU Tours, Tours
  - Hôpital Foch, Suresnes, Île-de-France Region
- Germany (10):
  - Universitätsmedizin Mannheim, Universität Heidelber, Mannheim, Baden-Wurttemberg
  - Klinikum Osnabrück GmbH, Osnabrück, Lower Saxony
  - Universitätsklinikum RWTH Aachen, Aachen, North Rhine-Westphalia
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel, Schleswig-Holstein
  - Universitätsklinikum Knappschaftskrankenhaus GmbH Bochum, Bochum
  - Universitätsklinikum Frankfurt, Frankfurt
  - Universitätsmedizin Göttingen, Göttingen
  - Medizinische Fakultät der Otto-von-Guericke-Universität Magdeburg, Magdeburg
  - Klinikum rechts der Isar der Technischen Universität München, München
  - Klinikum Vest GmbH, Recklinghausen
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitari Germans Trias i Pujol, Barcelona
- Switzerland (7):
  - Dept. of Neurology, Kantonsspital Aarau, Aarau, Canton of Aargau
  - Dept. of Neurology, Centre hospitalier universitaire vaudois (CHUV), Lausanne, Canton of Vaud
  - Dept. of Neurology, Ospedale Civo of Lugano, Lugano, Canton Ticino
  - Dept. of Neurology, Bern University Hospital, Bern
  - Hôpitaux Universitaires de Genève - HUG, Geneva
  - Kantonsspital St.Gallen, Sankt Gallen
  - Dept. of Neuroradiology, UniversitätsSpital Zürich, Zurich
- United Kingdom (3):
  - Belfast City Hospital, Belfast
  - St George's University Hospitals NHS Foundation Trust, London
  - Salford Royal, Salford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fladt J, Kaesmacher J, Meinel TR, Butikofer L, Strbian D, Eker OF, Albucher JF, Desal H, Marnat G, Papagiannaki C, Richard S, Requena M, Lapergue B, Pagano P, Ernst M, Wiesmann M, Boulanger M, Liebeskind DS, Gralla J, Fischer U. MRI vs CT for Baseline Imaging Evaluation in Acute Large Artery Ischemic Stroke: A Subanalysis of the SWIFT-DIRECT Trial. Neurology. 2024 Jan 23;102(2):e207922. doi: 10.1212/WNL.0000000000207922. Epub 2023 Dec 14. PMID 38165324
- [Derived] Mujanovic A, Eker O, Marnat G, Strbian D, Ijas P, Preterre C, Triquenot A, Albucher JF, Gauberti M, Weisenburger-Lile D, Ernst M, Nikoubashman O, Mpotsaris A, Gory B, Tuan Hua V, Ribo M, Liebeskind DS, Dobrocky T, Meinel TR, Buetikofer L, Gralla J, Fischer U, Kaesmacher J; SWIFT DIRECT investigators. Association of intravenous thrombolysis and pre-interventional reperfusion: a post hoc analysis of the SWIFT DIRECT trial. J Neurointerv Surg. 2023 Nov;15(e2):e232-e239. doi: 10.1136/jnis-2022-019585. Epub 2022 Nov 17. PMID 36396433
- [Derived] Meinel TR, Kaesmacher J, Buetikofer L, Strbian D, Eker OF, Cognard C, Mordasini P, Deppeler S, Mendes Pereira V, Albucher JF, Darcourt J, Bourcier R, Guillon B, Papagiannaki C, Costentin G, Sibolt G, Raty S, Gory B, Richard S, Liman J, Ernst M, Boulanger M, Barbier C, Mechtouff L, Zhang L, Marnat G, Sibon I, Nikoubashman O, Reich A, Consoli A, Weisenburger D, Requena M, Garcia-Tornel A, Saleme S, Moulin S, Pagano P, Saliou G, Carrera E, Janot K, Boix M, Pop R, Della Schiava L, Luft A, Piotin M, Gentric JC, Pikula A, Pfeilschifter W, Arnold M, Siddiqui A, Froehler MT, Furlan AJ, Chapot R, Wiesmann M, Machi P, Diener HC, Kulcsar Z, Bonati L, Bassetti C, Escalard S, Liebeskind D, Saver JL, Fischer U, Gralla J; SWIFT-DIRECT investigators. Time to treatment with bridging intravenous alteplase before endovascular treatment:subanalysis of the randomized controlled SWIFT-DIRECT trial. J Neurointerv Surg. 2023 Sep;15(e1):e102-e110. doi: 10.1136/jnis-2022-019207. Epub 2022 Jul 28. PMID 35902234
- [Derived] Fischer U, Kaesmacher J, Strbian D, Eker O, Cognard C, Plattner PS, Butikofer L, Mordasini P, Deppeler S, Pereira VM, Albucher JF, Darcourt J, Bourcier R, Benoit G, Papagiannaki C, Ozkul-Wermester O, Sibolt G, Tiainen M, Gory B, Richard S, Liman J, Ernst MS, Boulanger M, Barbier C, Mechtouff L, Zhang L, Marnat G, Sibon I, Nikoubashman O, Reich A, Consoli A, Lapergue B, Ribo M, Tomasello A, Saleme S, Macian F, Moulin S, Pagano P, Saliou G, Carrera E, Janot K, Hernandez-Perez M, Pop R, Schiava LD, Luft AR, Piotin M, Gentric JC, Pikula A, Pfeilschifter W, Arnold M, Siddiqui AH, Froehler MT, Furlan AJ, Chapot R, Wiesmann M, Machi P, Diener HC, Kulcsar Z, Bonati LH, Bassetti CL, Mazighi M, Liebeskind DS, Saver JL, Gralla J; SWIFT DIRECT Collaborators. Thrombectomy alone versus intravenous alteplase plus thrombectomy in patients with stroke: an open-label, blinded-outcome, randomised non-inferiority trial. Lancet. 2022 Jul 9;400(10346):104-115. doi: 10.1016/S0140-6736(22)00537-2. PMID 35810756
- [Derived] Fischer U, Kaesmacher J, S Plattner P, Butikofer L, Mordasini P, Deppeler S, Cognard C, Pereira VM, Siddiqui AH, Froehler MT, Furlan AJ, Chapot R, Strbian D, Wiesmann M, Bressan J, Lerch S, Liebeskind DS, Saver JL, Gralla J; SWIFT DIRECT study investigators. SWIFT DIRECT: Solitaire With the Intention For Thrombectomy Plus Intravenous t-PA Versus DIRECT Solitaire Stent-retriever Thrombectomy in Acute Anterior Circulation Stroke: Methodology of a randomized, controlled, multicentre study. Int J Stroke. 2022 Jul;17(6):698-705. doi: 10.1177/17474930211048768. Epub 2021 Oct 14. PMID 34569878